CLINICAL TRIAL: NCT03942718
Title: Internet-based Supervised Exercise Program in Systemic Lupus Erythematosus: A Randomized Controlled Trial
Brief Title: Systemic Lupus Erythematosus Exercise Program
Acronym: SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Mainz (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julia Weinmann-Menke, Head of the Department of Nephrology and Dialysis, University Medical Center Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniversityMedCntrMainz
Record Dates: First submitted 2019-01-25; First posted 2019-05-08 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Exercise; Aerobic training; Anaerobic training; Internet-based exercise program
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The three study arms (TAU, aerobic exercise, anerobic exercise) will be included in parallel. After 12 weeks, the patients in the control group will be invited to participate in the training group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Participants will obtain no exercise program. After 12 weeks, the patients in the control group will be invited to participate in the training group.
- Aerobic exercise group (Experimental): Participants will obtain aerobic exercise only.
  Interventions: Other: Exercise
- Anaerobic exercise group (Experimental): Participants will obtain aerobic and anaerobic exercise respectively
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will obtain an individualized exercise program based on entrance examination on treadmill.
  Arms: Aerobic exercise group; Anaerobic exercise group

SUMMARY:
This pilot study is a randomized controlled trial to assess the effect of an individualized supervised exercise program in patients with systemic lupus erythematosus (SLE) compared to treatment-as-usual (TAU).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of a 12-week individualized exercise program in subjects with SLE in comparison to treatment-as-usual therapy. Several previous studies showed that exercise leads to various benefits in treating SLE, including enhanced aerobic capacity, reduced symptoms of depression and fatigue. Moreover, it has been shown that exercise is well tolerated and does not impair disease activity in SLE negatively. Here, the effects of an individual internet-based exercise therapy for 12 weeks will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Positive ANA-titer (≥ 1:80) or Anti-dsDNA (≥ 200 IU/ml) or Highly avid-dsDNA autoantibody (≥ 30 IU/ml)
* Stable immunosuppressive therapy more than 30 days before beginning of the study with steroid (0-20 mg/day) or other immunosuppressive medication like Hydroxchloroquin, Chloroquin, Azathioprin, Methotrexat, Mycophenolatmofetil, Cyclosporin, Belimumab, Rituximab

Exclusion Criteria:

* Pregnancy, Active lupus nephritits, Physical activity more than two times a week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2peak) | 12-weeks
  Change of VO2peak after 12-weeks compared to baseline.

SECONDARY OUTCOMES:
Fatigue Scale for Motor and Cognitive Functions (FSMC) | 12-weeks
  Change of FSMC score after 12-weeks compared to baseline. The FSMC consists of 20 items (five-point Likert scale, from "absolutely agree" to "absolutely disagree") to assess cognitive fatigue (10 items) and motor fatigue (10 items). The summed scores for cognitive and motor fatigue result in the sum score. A cut-off value of 43 indicates mild fatigue, whereas higher values are associated with moderate fatigue (≥53) or severe fatigue (≥63).
Beck Depression Inventar (BDI) | 12-weeks
  Change of BDI score after 12-weeks compared to baseline to measure the severity of depression. The BDI questionnaire consists of 21 sets of statements. Each set consists of 4 statements which are ranked in terms of severity from 0 to 3. The sum of the item scores (range 0-63) indicates the severity of depression. The standardized scale is: 0-8: no depression. 9-13: minimal depression. 14-19: mild depression. 20-28: moderate depression. 29-63: severe depression.
Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) | 12-weeks
  The Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) - Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) (SELENA-SLEDAI) will be used to measure the disease activity. The index consist of 24 items including clinical and laboratory variables to measure disease activity within the previous 10 days. The maximum score is 105. SLEDAI scores >3 indicate a mild or moderate flare, SLEDAI ≥12 indicate a severe flare.
Disease Activity Score 28 (DAS 28) | 12-weeks
  Change of DAS 28 score after 12-weeks compared to baseline. The DAS 28 score indicates rheumatoid arthritis disease activity and treatment response. The score composes of 4 measures including the number of swollen/tender joints, C reactive protein and patients health assessment. A total score is calculated using the DAS 28 formula. Values range from 2.0 to 10, whereas higher values indicate higher disease activity.
Work Ability Index (WAI) | 12-weeks
  The WAI self-assessment questionnaire will be used to assess the workability of the patients. The questionnaire covers six dimensions including current workability, as well as past 2 year estimation among others. The answers have different scores, which are summed to a total score, leading to four categories. 7-27 points indicate bad, 28-36 points moderate, 37-43 good, and 44-49 points very good workability.
Circulating, cell-free Deoxyribonucleic acid (CfDNA) | 12-weeks
  The concentration of cfDNA (ng/ml) will be measured during and after acute exercise at baseline and after 12-weeks exercise intervention using quantitative PCR. Compared to healthy subjects SLE patients show higher cfDNA plasma levels.
Revised Cutaneous Lupus Erythematosus Disease Area and Severity Index (RCLASI) | 12-weeks
  Change of score on RCLASI after 12-weeks compared to baseline. The RCLASI scoring system includes the RCLASI Activity Score to measure the activity of skin lesions, and the RCLASE Damage Score to measure the damage of skin lesions in patients with discoid lupus erythematosus and cutaneous lupus erythematosus. The score is used as a follow-up parameter for the Lupus activity of the skin. It was also shown that RCLASI correlates well with the physicians and patients global assessment of disease activity.
Extra cellular vesicles (EVs) | 12-weeks
  The relative amount of EV subpopulations will be analyzed before and after acute exercise, as well as after 12-weeks of exercise intervention using bead isolation and or size exclusion chromatography followed by protein marker characterization.
Autoantibodies | 12-weeks
  Change of antinuclear antibodies (ANA) titer after 12-weeks of exercise intervention compared to baseline (standard value ≤1:80).
Ventilatory threshold (VT) | 12-weeks
  Change of VT after 12-weeks compared to baseline.
Muscle mass | 12-weeks
  Change of muscle mass after 12-weeks compared to baseline. Muscle mass will be measured in absolute mass [kg] including internal organs using bioelectrical impedance analysis (InBody 3.0 Body composition analyzer).
Chair-Stand-Test (CST) | 12-weeks
  Change of CST after 12-weeks compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Weinmann-Menke, Prof. Dr. med, Study Director — University mainz, Center of medicine
Locations (1):
- UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz I. Medizinische Klinik und Poliklinik, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Pisareva E, Mihalovicova L, Pastor B, Kudriavtsev A, Mirandola A, Mazard T, Badiou S, Maus U, Ostermann L, Weinmann-Menke J, Neuberger EWI, Simon P, Thierry AR. Neutrophil extracellular traps have auto-catabolic activity and produce mononucleosome-associated circulating DNA. Genome Med. 2022 Nov 28;14(1):135. doi: 10.1186/s13073-022-01125-8. PMID 36443816
- [Derived] Boedecker SC, Philippi KFA, Neuberger E, Schmidt S, Pfirrmann D, Haller N, Schwarting A, Simon P, Weinmann-Menke J. Twelve-Week Internet-Based Individualized Exercise Program in Adults With Systemic Lupus Erythematosus: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Nov 3;9(11):e18291. doi: 10.2196/18291. PMID 33141101